CLINICAL TRIAL: NCT02831582
Title: Prevention of Aromatase Inhibitor-Induced Toxicity With Omega-3 Supplementation
Brief Title: Omega-3 Supplementation in Prevention of Aromatase Inhibitor-Induced Toxicity in Patients With Stage I-III Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Nicole Williams, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OSU-15222; NCI-2016-00377 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2016-05-01; First posted 2016-07-13 (Estimated); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Arthralgia; Breast Neoplasms
Keywords: Breast Cancer; Postmenopausal; Stage IA; Stage IB; Stage IIA; Stage IIB; Stage IIIA; Stage IIIB; Stage IIIC
MeSH Terms: conditions — Arthralgia; Breast Neoplasms | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (omega-3 fatty acid) (Active Comparator): Patients receive omega-3 fatty acid supplementation PO QD for 6 months.
  Interventions: Dietary Supplement: Omega-3 Fatty Acid
- Arm II (placebo) (Placebo Comparator): Patients receive placebo PO QD for 6 months.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acid — Given PO.
  Other Names: n-3 Fatty Acid; Omega 3 Fatty Acid; OMEGA-3 FATTY ACIDS; Omega-3 Polyunsaturated Fatty Acid; Omega-3 PUFA; omega-3-Fatty Acids
  Arms: Arm I (omega-3 fatty acid)
Other: Placebo — Given PO.
  Other Names: placebo therapy; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This clinical trial studies the use of omega-3 fatty acid supplementation in preventing aromatase inhibitor-induced toxicity in patients with stage I-III breast cancer. An omega-3 supplementation may help relieve moderate to severe bone pain and improve joint symptoms caused by aromatase inhibitor-induced arthralgias.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of the complementary therapy omega-3 fatty acid (n-3 PUFA) supplementation in preventing aromatase inhibitor-induced arthralgias (AIIAs).

SECONDARY OBJECTIVES:

I. To prospectively define the population most at risk for developing AIIAs by the identification and validation of genetic risk predictors and to develop a single nucleotide polymorphism (SNP)/gene profile predictive of treatment intervention response.

OUTLINE: Patients are randomized to 1 of 2 groups.

Group I: Patients receive omega-3 fatty acid supplementation orally (PO) once daily (QD) for 6 months.

Group II: Patients receive placebo PO QD for 6 months.

After completion of study, patients will be followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with breast cancer stages I-III initiating first line adjuvant aromatase inhibitor (AI) therapy with any of the FDA-approved AIs (anastrazole, exemestane, letrozole)
* Concurrent gonadotropin-releasing hormone (GnRH) agonist therapy is allowed; concurrent breast related radiation therapy is allowed.
* Prior tamoxifen use is allowed
* Prior chemotherapy is allowed
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Metastatic malignancy of any kind
* Rheumatoid arthritis and other types of autoimmune and inflammatory joint disease
* AI use > 21 days prior to study enrollment
* Known bleeding disorders
* Current use of warfarin or other anticoagulants
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situation that would limit compliance with study requirements
* Daily use of n-3 PUFA concentrates or capsules or any other supplements that might interact with n-3 PUFA supplements if > 375 mg per day of of eicosapentaenoic acid (EPA)/ docosahexaenoic acid (DHA) within six months of study initiation
* Pregnant or nursing women
* Known sensitivity or allergy to fish or fish oil
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2016-10-12 (Actual); Primary Completion 2021-12-11 (Actual); Study Completion 2021-12-11 (Actual)

PRIMARY OUTCOMES:
Change in pain score based on the Brief Pain Inventory (BPI) | Baseline to up to 6 months
  Analysis of patterns of change over time in pain scores through the application of hierarchical linear regression models.

SECONDARY OUTCOMES:
Change in joint symptoms based on quality of life instruments | Baseline to up to 6 months
  An exploratory analysis, logistic mixed effect regression models will be used to compare the occurrence of moderate to severe joint symptoms during the 6 month period between the two treatment groups.
Change in joint symptoms based on symptomatology instruments | Baseline to up to 6 months
  An exploratory analysis, logistic mixed effect regression models will be used to compare the occurrence of moderate to severe joint symptoms during the 6 month period between the two treatment groups.
Identification and validation of genetic risk predictors for aromatase inhibitor-induced arthralgias | Up to 6 months
  Interaction tests between treatment and stratification variables will be conducted to explore whether these factors are predictive of average pain scores.
Rate of compliance | Up to 6 months
  The rates of adherence to and discontinuation of AI therapy will be recorded. Reasons for treatment discontinuation will be described. In addition, the investigators will also examine the compliance rates with n-3 PUFA or placebo supplements with pill counts at each visit and with a patient recorded medication calendar.
SNP analysis by standard data preprocessing operations and sequential analysis | Up to 6 months
  A sequential analysis of the data that allows filtering of extraneous SNPs and select SNP loci, identification and creation of predictive SNP clusters, and then evaluation of the networks' potential clinical and biological validity will be performed.

OTHER OUTCOMES:
Level of inflammatory markers | Up to 6 months
Red blood cells (RBC) n-3 PUFA levels | Up to 6 months
  The relationship between RBC n-3 PUFA levels, inflammatory blood markers and the joint symptoms evaluated by the patient symptom assessment instruments. Scatter plots and correlation coefficients (either Pearson or Spearman) will be used to summarize their pairwise relation. The differences between the treatment and placebo in terms of these measures will also be reported using numerical summaries and graphic plots.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Williams, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Cleveland Clinic Cancer Center/Fairview Hospital, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts KE, Adsett IT, Rickett K, Conroy SM, Chatfield MD, Woodward NE. Systemic therapies for preventing or treating aromatase inhibitor-induced musculoskeletal symptoms in early breast cancer. Cochrane Database Syst Rev. 2022 Jan 10;1(1):CD013167. doi: 10.1002/14651858.CD013167.pub2. PMID 35005781
- See also: The Jamesline — http://cancer.osu.edu